CLINICAL TRIAL: NCT01397318
Title: Effects of Modified TaiChi Exercise on Maternal Stress, Fatigue, Sleep Quality, Biomarkers, and Infant Gestational Age and Birthweight
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Szu-Yuan Chou, Department of Obsterics & Gynecology, WanFang Hospital
Other Study IDs: 100005
Record Dates: First submitted 2011-07-15; First posted 2011-07-19 (Estimated); Last update posted 2011-07-19 (Estimated); Status verified 2011-07

CONDITIONS: TaiChi Exercise; Pregnant Women
Keywords: TaiChi Exercise; pregnant women

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Experimental Group
- Control Group

SUMMARY:
Many pregnant women experience stress, fatigue, and poor sleep quality that may influence infant outcomes such as prematurity and low birthweight through immunologic pathway of biomarkers (serum cytokines and c-reactive protein). In contrast, TaiChi exercise, one kind of physical activity, can increase pulmonary and immune functions and reduce stress may therefore prevent pregnancy complications and further prevent adverse pregnancy outcomes; however, its effects has not been explored in studies. Therefore, this study aims to investigate relationships between prenatal stress, fatigue, sleep quality, biomarkers, and infant outcomes; modified a TaiChi exercise program suitable for pregnant women; and test the effects of the exercise on reducing stress and fatigue, promote sleep quality, modulate biomarkers, and prevent adverse infant outcomes. Infant outcomes in the study will be measured with gestational age and birthweight. The study is a three-stage longitudinal interventional design.

DETAILED DESCRIPTION:
In the first-stage, patterns of prenatal stress, fatigue, and sleep quality will be investigated by surveying 300 pregnant women who are over 23 weeks of gestation and screen for pregnant women with fatigue and poor sleep quality. In the second-stage, experts in obstetrics and TaiChi will be invited to modify a TaiChi exercise program. Thirty women who experience fatigue and poor sleep quality will be invited to practice the modified TaiChi exercise. Comments from those participants on the program will be used to refine the program and a DVD will be made. After the program is well-designed and recorded, participants recruited for the third-stage study will be randomly assigned to TaiChi or comparison group. They will be asked to complete questionnaires and give blood samples for biomarker tests when they are at 27-29, 31-33, and 35-37 weeks of gestation; in labor; and at 4-6 weeks postpartum. In addition to practice the exercise at home, participants in the TaiChi group will practice TaiChi in groups every month. In contrast, comparison group will be asked to keep on their usual daily activities, no other interventions will be introduced. Phone calls or postcard will be made or sent routinely to participants to ensure their long-term participation. Questionnaires used for the study include 10-item Perceived Stress Scale, Multidimensional Assessment of Fatigue Scale, and Pittsburgh Sleep Quality Index. Descriptive statistics, Pearson correlation, and generalized estimating equations will be applied to understand predictive effects of maternal stress, fatigue, sleep quality, and biomarkers on infant outcomes; and effects of modified TaiChi exercise on maternal stress, fatigue, sleep quality, biomarkers, and infant outcomes. In addition to develop a modified TaiChi exercise program suitable for pregnant women, the study anticipates that maternal stress, fatigue, and poor sleep quality can predict infant outcomes through immunologic pathway, and the modified TaiChi exercise can reduce maternal stress and fatigue, improve sleep quality, modulate biomarkers, and hence prevent adverse infant outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Criteria for participation are women who:

  * are over 17;
  * can read Chinese;
  * are at or over 24 weeks of gestation;
  * pregnant with singleton;
  * are not diagnosed of pregnancy complications such as preeclampsia, preterm labor, preterm rupture of membranes, gestational diabetes, and cervical incompetence before recruitment; and
  * are willing to complete questionnaires and give blood samples.

Exclusion Criteria:

* pregnant women who do not meet the recruitment criteria will be excluded from the study.

Min Age: 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: pregnant women
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2010-09; Study Completion 2013-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Szu-Yuan Chou, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University-WanFang Hospital, Taipei, Taiwan